CLINICAL TRIAL: NCT04267770
Title: A Study of Flat and Circadian Insulin Infusion Rates in Continuous Subcutaneous Insulin Infusion (CSII) in Adults With Type 1 Diabetes
Brief Title: Flat and Circadian Insulin Infusion Rates in Continuous Subcutaneous Insulin Infusion
Acronym: FIRST1D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17HH4255
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Results first posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- circadian insulin infusion rates (Experimental): Initial variable basal rates aim to replicate circadian changes in insulin requirements and are derived from total basal insulin in adults over 24 years old, and from weight in adults aged 18 to 24 years.
  Interventions: Drug: Insulin (circadian)
- flat rates (Active Comparator): flat basal rate
  Interventions: Drug: Insulin (flat rate)

INTERVENTIONS:
Drug: Insulin (circadian) — Participant's own insulin adjusted to circadian infusion rates
  Arms: circadian insulin infusion rates
Drug: Insulin (flat rate) — Participant's own insulin set to flat basal rates
  Arms: flat rates

SUMMARY:
Randomised controlled trial to contribute to the evidence base for the optimal initial insulin profile for adults with type 1 diabetes commencing insulin pump therapy.

DETAILED DESCRIPTION:
Initiation of insulin pump therapy in people with type 1 diabetes requires conversion of a basal insulin dose, given as once or twice daily long-acting insulin, to a continuous basal infusion regimen. This conversion may be based on basal insulin dose only, or total daily insulin dose, and may result in a flat basal insulin profile or an initial variable basal rate.

Initial variable basal rates aim to replicate circadian changes in insulin requirements and are derived from total basal insulin in adults over 24 years old, and from weight in adults aged 18 to 24 years. Initial rates were developed from 63 well-controlled people with type 1 diabetes over 14 years of age and have been assessed against a flat basal rate in a small randomised controlled trial with 12 participants. Mean glucose was lower in the circadian basal rate group with particular differences noted in the early morning when glucose rises were more pronounced in the flat basal rate group1.

In 50 people with type 1 diabetes treated with insulin pump therapy, HbA1c was lower in those with lower basal rates at midnight, and in those with higher basal rates in the afternoon, suggesting a benefit of circadian patterns2. In 33 people with type 1 diabetes over 16 years of age basal rate distribution established at commencement of pump therapy did not alter over 6 months3. However, a 6 month cross-over study of circadian rates and oligophasic basal rates showed no difference in HbA1c4.

Following initiation on insulin pump therapy basal rates are personalised to capillary blood and continuous interstitial fluid glucose monitoring.

In adults with type 1 diabetes starting insulin pump therapy there are limited data to guide the optimal insulin profile to rapidly achieve target glucose and minimise healthcare professional input.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age
* Diagnosis of T1DM for > 1 year
* On MDI with decision made to commence CSII
* Structured education in previous 3 years
* HbA1c ≤ 75mmol/mol (9%)
* Stimulated c-peptide <200pmol/L
* No severe hypoglycaemia (defined as needing 3rd party assistance) in previous year

Exclusion Criteria:

* Previous CSII
* Night or shift worker
* Recurrent severe hypoglycaemia
* Pregnant or planning pregnancy
* Breastfeeding
* Enrolled in other clinical trials
* Have active malignancy or under investigation for malignancy
* Addison's Disease
* Gastroparesis
* Autonomic neuropathy
* Concomitant use of GLP-1 analogues and gliptins
* Visual impairment
* Reduced manual dexterity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2018-11-09 (Actual); Study Completion 2018-11-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College Clinical Research Facility, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Circadian Insulin Infusion Rates | Flat Rates
Started | 9 | 8
Completed | 9 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Circadian Insulin Infusion Rates | Flat Rates | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.3 (8.6) | 33.3 (8.6) | 33.3 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 11
  Male | 1 | 5 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Basal Insulin Rate
Description: Absolute change in insulin basal rate over 24 hours after 3 rounds of basal rate testing (calculated by the sum of absolute changes for each 1 hour block compared with baseline)
Time Frame: over 24 hours after 3 rounds of basal rate testing
Measure: Median (Inter-Quartile Range); unit: Units of insulin
Arm/Group | Circadian Insulin Infusion Rates | Flat Rates
Number analyzed (Participants) | 9 | 8
Units of insulin | 1.8 [0.63 to 2.99] | 1.49 [0.83 to 1.94]

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Circadian Insulin Infusion Rates | Flat Rates
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 0/9 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-23): https://cdn.clinicaltrials.gov/large-docs/70/NCT04267770/Prot_SAP_000.pdf